CLINICAL TRIAL: NCT05597085
Title: A Retrospective Analysis of Inotuzumab Ozogamicin (InO) Usage in Adult Patients With Relapsed/Refractory (R/R) B-cell Acute Lymphoblastic Leukemia (ALL)
Brief Title: A Study of Patients Who Received Inotuzumab Ozogamicin for B-cell ALL (Acute Lymphoblastic Leukemia) That Occurred Again After the Last Treatment
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1931043; NCT05597085 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Adult Relapsed/Refractory B Cell Acute Lymphoblastic Leukemia
Keywords: Relapsed ALL; Refractory ALL; Adult Relapsed/Refractory ALL; Adult ALL; Relapsed B Cell ALL; Refractory B Cell ALL; Relapsed Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Adult relapsed or refractory B Cell ALL: Adult patients whose B Cell ALL has occurred again after the last treatment or patients who never responded to prior treatment
  Interventions: Drug: Inotuzumab Ozogamicin

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin — Inotuzumab Ozogamicin is an Antibody drug conjugate directed against CD 22 positive B Cell ALL
  Other Names: Besponsa; Inonza

SUMMARY:
The purpose of the study was to understand the effectiveness and safety of the study medicine called Inotuzumab ozogamicin (InO) in patients with B-cell ALL in whom the disease occurred again after the last treatment.

This retrospective Study enroll adult patients who:

* were CD22 positive (a molecule in the body that stops the over activity of the immune system)
* Received only InO for the treatment of B-cell ALL that occurred again after the last treatment
* were Philadelphia chromosome positive (which occurs because of changes in genes)
* failed treatment with at least one Tyrosine Kinase Inhibitor (type of medicine that blocks the action of enzymes called tyrosine kinases which takes care of many cell functions, such as cell growth and division).

The patient data except their personal details are collected from a hospital based electronic medical record in India.

In this study the effectiveness and safety of InO will be studied after it was released to the market.

To do that, the study aims to gather details of B-cell ALL patients from 7 -10 hospitals across India:

* in whom the disease occurred again
* or those who never showed any improvement to earlier treatments
* now being treated with InO alone

Around 55 patients who have taken InO are likely to be enrolled in the study.

Then by using a statistical model and with all the information gathered, the safety and effectiveness of InO will be decided.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years old at the initiation of InO treatment

  * Patients with relapsed/refractory B-cell ALL
  * Patients who initiated InO monotherapy between Feb'2017 and Feb'2022 and are CD22 positive
  * Ph+ patients who have failed treatment with at least 1 TKI

Exclusion Criteria:

* Patient not completing at least 1 cycle of InO therapy • Patient on InO in combination with chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Relapsed or Refractory B Cell Acute Lymphoblastic Leukemia Patients
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- India (5):
  - Fortis Memorial Research Institute, Gurugram, Haryana
  - Malabar Cancer Center, Thalassery, Kerala
  - Rajiv Gandhi Cancer Institute and Research Centre, New Delhi, National Capital Territory of Delhi
  - Indo-American Cancer & Research Centre, Hyderabad, Telangana
  - Tata Medical Center, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1931043

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of eligible Indian participants with Relapsed/Refractory/ B Cell Acute lymphoblastic leukemia (R/R B cell ALL), who aged greater than or equal to 18 years at the time of initiating treatment with Inotuzumab ozogamicin (InO) [index date], was collected retrospectively from hospital medical records. For eligibility Index date could have been between Feb 2017 to Feb 2022. Available data was retrieved from 08-Mar-2023 to 10-Jul-2023 (approximately 4 months) in the current observational study.
Groups:
- Inotuzumab Ozogamicin (InO): Participants who were treated with InO as a monotherapy and completed at least one cycle of InO and were CD22 positive, in real world setting under routine clinical practice outside of clinical trials were observed retrospectively.
Period: Overall Study
Arm/Group | Inotuzumab Ozogamicin (InO)
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants whose data was retrieved and observed in the study.
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Age, Customized [Count of Participants; unit: Participants]
  18-50 years | 23
  Above (>) 50 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Complete Remission (CR) or Complete Remission With Incomplete Hematological Recovery (CRi) Following Treatment With InO
Description: CR was defined as 5 percent (%) bone marrow blasts, no evidence of disease in the bone marrow, and recovery of peripheral blood count (platelet count of [more than] >100*10^9 cells/liter [L] and absolute neutrophil count of >1*10^9 cells/L). CRi was defined as 5% bone marrow blasts and no evidence of disease in the bone marrow, but with incomplete recovery of peripheral blood count.
Time Frame: From InO treatment initiation (Apr 2018) till end of follow-up (Apr 2023) [Maximum up to 61 Months]; data retrospectively collected from 08-Mar-2023 to 10-Jul-2023 (approximately 4 months of this study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Participants | 19

2. Primary Outcome: Number of Participants Who Achieved Complete Remission (CR) or Complete Remission With Incomplete Hematological Recovery (CRi) Following Treatment With InO, Classified Per Number of Lines of Salvage Therapies Prior to InO Initiation
Description: CR was defined as 5 percent (%) bone marrow blasts, no evidence of disease in the bone marrow, and recovery of peripheral blood count (platelet count of [more than] >100*10^9 cells/liter [L] and absolute neutrophil count of >1*10^9 cells/L). CRi was defined as 5% bone marrow blasts and no evidence of disease in the bone marrow, but with incomplete recovery of peripheral blood count. Salvage therapy is use of drugs after standard conventional chemotherapeutic regimens have failed to achieve remission.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Participants
  Participants achieved CR/CRi during first salvage therapy: number analyzed (Participants) | 10
  Participants achieved CR/CRi during first salvage therapy | 6
  Participants achieved CR/CRi during second salvage therapy: number analyzed (Participants) | 18
  Participants achieved CR/CRi during second salvage therapy | 11
  Participants achieved CR/CRi during third salvage therapy: number analyzed (Participants) | 4
  Participants achieved CR/CRi during third salvage therapy | 2

3. Primary Outcome: Number of Participants Who Achieved CR or CRi Following Treatment With InO, Classified Per High Burden and Low Burden Disease
Description: CR was defined as 5% bone marrow blasts, no evidence of disease in the bone marrow, and recovery of peripheral blood count (platelet count of >100*10^9 cells/L and absolute neutrophil count of >1*10^9 cells/L). CRi was defined as 5% bone marrow blasts and no evidence of disease in the bone marrow, but with incomplete recovery of peripheral blood count. Disease burden was defined using percentage of bone marrow blasts (BMB). In this outcome measure low disease burden indicated BMB <50% and high disease burden indicated BMB >=50%.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Participants
  Participants achieved CR/CRi: BMB <50%: number analyzed (Participants) | 16
  Participants achieved CR/CRi: BMB <50% | 10
  Participants achieved CR/CRi: BMB >=50%: number analyzed (Participants) | 16
  Participants achieved CR/CRi: BMB >=50% | 9

4. Secondary Outcome: Number of Participants Who Achieved Minimal Residual Disease (MRD) Negativity Following Initiation of Ino Among Those Who Had CR/CRi
Description: Negative MRD was defined as documented in medical records or (if unavailable in the records) as leukemic cells comprising <1*10^-4 (<0.01%) of bone marrow nucleated cells. MRD was assessed by multicolor flow cytometry. CR was defined as 5% bone marrow blasts, no evidence of disease in the bone marrow, and recovery of peripheral blood count (platelet count of >100*10^9/L and absolute neutrophil count of >1*10^9/L). CRi was defined as 5% bone marrow blasts and no evidence of disease in the bone marrow, but with incomplete recovery of peripheral blood count.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 19
Participants
  Participants with CR who achieved MRD: number analyzed (Participants) | 18
  Participants with CR who achieved MRD | 17
  Participants with CRi who achieved MRD: number analyzed (Participants) | 1
  Participants with CRi who achieved MRD | 1

5. Secondary Outcome: Number of Participants Who Achieved MRD Negativity Classified Per Number of Lines of Salvage Therapies Following Initiation of InO Among Those Who Had CR/CRi
Description: Negative MRD was defined as documented in medical records or (if unavailable in the records) as leukemic cells comprising <1*10^-4 (<0.01%) of bone marrow nucleated cells. MRD was assessed by multicolour flow cytometry. CR was defined as 5% bone marrow blasts, no evidence of disease in the bone marrow, and recovery of peripheral blood count (platelet count of >100*10^9/L and absolute neutrophil count of >1*10^9/L). CRi was defined as 5% bone marrow blasts and no evidence of disease in the bone marrow, but with incomplete recovery of peripheral blood count. Salvage therapy is use of drugs after standard conventional chemotherapeutic regimens have failed to achieve remission. Participants with either CR or CRi who achieved MRD negativity classified per number of lines of salvage therapies are reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 19
Participants
  First Salvage Therapy: number analyzed (Participants) | 6
  First Salvage Therapy | 5
  Second Salvage Therapy: number analyzed (Participants) | 11
  Second Salvage Therapy | 11
  Third Salvage Therapy: number analyzed (Participants) | 2
  Third Salvage Therapy | 2

6. Secondary Outcome: Number of Participants Who Achieved MRD Negativity Classified Per High Burden and Low Burden Disease Following Initiation of InO Among Those Who Had CR/CRi
Description: Negative MRD was defined as documented in medical records or (if unavailable in the records) as leukemic cells comprising <1*10^-4 (<0.01%) of bone marrow nucleated cells. MRD was assessed by multicolour flow cytometry. CR was defined as 5% bone marrow blasts, no evidence of disease in the bone marrow, and recovery of peripheral blood count (platelet count of >100*10^9/L and absolute neutrophil count of >1*10^9/L). CRi was defined as 5% bone marrow blasts and no evidence of disease in the bone marrow, but with incomplete recovery of peripheral blood count. Disease burden was defined using percentage of BMB. In this outcome measure low disease burden indicated BMB <50% and high disease burden indicated BMB >=50%. Participants with either CR or CRi who achieved MRD negativity classified per high burden and low burden disease are reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 19
Participants
  BMB <50%: number analyzed (Participants) | 10
  BMB <50% | 10
  BMB >=50%: number analyzed (Participants) | 9
  BMB >=50% | 8

7. Secondary Outcome: Number of Participants Achieving MRD Negativity Following Initiation of InO Among Those Who Had CR/CRi in Elderly Participants (>65 Years)
Description: Negative MRD was defined as documented in medical records or (if unavailable in the records) as leukemic cells comprising <1*10^-4 (<0.01%) of bone marrow nucleated cells. MRD was assessed by multicolour flow cytometry. CR was defined as 5% bone marrow blasts, no evidence of disease in the bone marrow, and recovery of peripheral blood count (platelet count of >100*10^9/L and absolute neutrophil count of >1*10^9/L). CRi was defined as 5% bone marrow blasts and no evidence of disease in the bone marrow, but with incomplete recovery of peripheral blood count.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 2
Participants | 2

8. Secondary Outcome: Median Number of Cycles of InO Treatment
Description: The median number of cycles of InO a participant received during treatment were included. Standard dose of InO: 1.8 mg/m^2 per 21 days cycle.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (Full Range); unit: Cycles of InO Treatment
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Cycles of InO Treatment | 2 [1 to 6]

9. Secondary Outcome: Median Number of Cycles of InO Needed to Attain CR/CRi
Description: CR was defined as 5% bone marrow blasts, no evidence of disease in the bone marrow, and recovery of peripheral blood count (platelet count of >100*10^9/L and absolute neutrophil count of >1*10^9/L). CRi was defined as 5% bone marrow blasts and no evidence of disease in the bone marrow, but with incomplete recovery of peripheral blood count.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. 'Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Cycles of InO treatment
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 19
Cycles of InO treatment | 2 [1 to 6]

10. Secondary Outcome: Mean Number of Cycles of InO Needed to Attain CR or CRi Classified Per Number of Lines of Salvage Therapies
Description: CR was defined as 5% bone marrow blasts, no evidence of disease in the bone marrow, and recovery of peripheral blood count (platelet count of >100*10^9/L and absolute neutrophil count of >1*10^9/L). CRi was defined as 5% bone marrow blasts and no evidence of disease in the bone marrow, but with incomplete recovery of peripheral blood count. Salvage therapy is use of drugs after standard conventional chemotherapeutic regimens have failed to achieve remission.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Cycles of InO treatment
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 19
Cycles of InO treatment
  First Salvage Therapy: number analyzed (Participants) | 6
  First Salvage Therapy | 2.33 (1.21)
  Second Salvage Therapy: number analyzed (Participants) | 11
  Second Salvage Therapy | 2.00 (1.48)
  Third Salvage Therapy: number analyzed (Participants) | 2
  Third Salvage Therapy | 3.50 (3.54)

11. Secondary Outcome: Duration of Remission (DOR)
Description: Remission was defined as either the reduction or disappearance of the signs and symptoms of leukemia for this study.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 17
Months | 6 [0.5 to 61]

12. Secondary Outcome: Number of Participants Categorized as Per InO Doses
Description: Standard dose of InO was 1.8 milligrams (mg) per meter square (m^2) per cycle. Under dose of InO was less than 1.8 mg/m^2 per cycle. Overdose of InO was more than 1.8 mg/m^2 per cycle.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Participants
  Under Dose | 17
  Standard Dose | 12
  Overdose | 3

13. Secondary Outcome: Number of Participants With InO Dose Modifications
Description: Number of participants for whom there was deviation in InO dose from the standard dose (1.8 mg/ m^2 per cycle) were included.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Participants
  Below standard dose | 17
  Above standard dose | 3

14. Secondary Outcome: Number of Participants Who Received Concomitant Medications
Description: Concomitant medication was defined as any medication other than, and in addition to, the study medication taken for any period of time during the treatment.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Participants | 0

15. Secondary Outcome: Number of Participants Who Proceeded to Hematopoietic Stem Cell Transplantation (HSCT)
Description: HSCT is the transplantation of multipotent hematopoietic stem cells to treat some type of cancers and other diseases.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Participants | 11

16. Secondary Outcome: Survival Rate at 6 and 12 Months in Transplanted and Non-Transplanted Participants Who Achieved CR/CRi and MRD Negativity
Description: Survival rate: percentage of participants in a study or treatment group who were still alive for a certain period of time after they were diagnosed with or started treatment for a disease. Negative MRD was defined as documented in medical records or (if unavailable in the records) as leukemic cells comprising <1*10^-4 (<0.01%) of bone marrow nucleated cells. MRD was assessed by multicolour flow cytometry. CR was defined as 5% bone marrow blasts, no evidence of disease in the bone marrow, and recovery of peripheral blood count (platelet count of >100*10^9 cells/L and absolute neutrophil count of >1*10^9 cells/L). CRi was defined as 5% bone marrow blasts and no evidence of disease in the bone marrow, but with incomplete recovery of peripheral blood count. In this outcome measure percentage of participants who had either CR or CRi with MRD negativity and survived at the end of 6 months and 12 months post initiation of InO treatment are reported on the basis of transplantation status.
Time Frame: 6 and 12 months post initiation of InO treatment; data retrospectively collected from 08-Mar-2023 to 10-Jul-2023 (approximately 4 months of this study)
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 18
Percentage of participants
  Transplanted Participants: Survival rate at 6 Months: number analyzed (Participants) | 9
  Transplanted Participants: Survival rate at 6 Months | 66.7
  Non-transplanted Participants: Survival rate at 6 Months: number analyzed (Participants) | 9
  Non-transplanted Participants: Survival rate at 6 Months | 88.9
  Transplanted Participants: Survival rate at 12 Months: number analyzed (Participants) | 9
  Transplanted Participants: Survival rate at 12 Months | 33.3
  Non-transplanted Participants: Survival rate at 12 Months: number analyzed (Participants) | 9
  Non-transplanted Participants: Survival rate at 12 Months | 44.4

17. Secondary Outcome: Survival Rate at 6 and 12 Months in Transplanted and Non-Transplanted Participants Classified Per Number of Lines of Salvage Therapies
Description: Survival rate was defined as the percentage of participants in a study or treatment group who were still alive for a certain period of time after they were diagnosed with or started treatment for a disease. Salvage therapy is use of drugs after standard conventional chemotherapeutic regimens have failed to achieve remission. In this outcome measure percentage of transplanted and non-transplanted participants who survived at the end of 6 months and 12 months post initiation of InO treatment are classified based on number of lines of salvage therapies.
Time Frame: as for outcome 16
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 30
Percentage of participants
  Transplanted participants: first salvage therapy: Survival rate at 6 months: number analyzed (Participants) | 0
  Transplanted participants: second salvage therapy: Survival rate at 6 months: number analyzed (Participants) | 9
  Transplanted participants: second salvage therapy: Survival rate at 6 months | 66.7
  Transplanted participants: third salvage therapy: Survival rate at 6 months: number analyzed (Participants) | 2
  Transplanted participants: third salvage therapy: Survival rate at 6 months | 50
  Transplanted participants: first salvage therapy: Survival rate at 12 months: number analyzed (Participants) | 0
  Transplanted participants: second salvage therapy: Survival rate at 12 months: number analyzed (Participants) | 9
  Transplanted participants: second salvage therapy: Survival rate at 12 months | 33.3
  Transplanted participants: third salvage therapy: Survival rate at 12 months: number analyzed (Participants) | 2
  Transplanted participants: third salvage therapy: Survival rate at 12 months | 50
  Non-transplanted participants: first salvage therapy: Survival rate at 6 months: number analyzed (Participants) | 9
  Non-transplanted participants: first salvage therapy: Survival rate at 6 months | 56
  Non-transplanted participants: second salvage therapy: Survival rate at 6 months: number analyzed (Participants) | 8
  Non-transplanted participants: second salvage therapy: Survival rate at 6 months | 25.0
  Non-transplanted participants: third salvage therapy: Survival rate at 6 months: number analyzed (Participants) | 2
  Non-transplanted participants: third salvage therapy: Survival rate at 6 months | 50
  Non-transplanted participants: first salvage therapy: Survival rate at 12 months: number analyzed (Participants) | 9
  Non-transplanted participants: first salvage therapy: Survival rate at 12 months | 33
  Non-transplanted participants: second salvage therapy: Survival rate at 12 months: number analyzed (Participants) | 8
  Non-transplanted participants: second salvage therapy: Survival rate at 12 months | 12.5
  Non-transplanted participants: third salvage therapy: Survival rate at 12 months: number analyzed (Participants) | 2
  Non-transplanted participants: third salvage therapy: Survival rate at 12 months | 50

18. Secondary Outcome: Survival Rate at 6 and 12 Months in Transplanted and Non-Transplanted Participants Classified Per High Burden and Low Burden Disease
Description: Survival rate was defined as the percentage of participants in a study or treatment group who were still alive for a certain period of time after they were diagnosed with or started treatment for a disease. Disease burden was defined using percentage of BMB. In this outcome measure low disease burden indicated BMB <50% and high disease burden indicated BMB >=50%. In this outcome measure percentage of transplanted and non-transplanted participants who survived at the end of 6 months and 12 months post initiation of InO treatment are classified based on high burden and low burden disease.
Time Frame: as for outcome 16
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 30
Percentage of participants
  Transplanted: BMB <50%: Survival rate at 6 Months: number analyzed (Participants) | 7
  Transplanted: BMB <50%: Survival rate at 6 Months | 71.43
  Transplanted: BMB >=50%: Survival rate at 6 Months: number analyzed (Participants) | 4
  Transplanted: BMB >=50%: Survival rate at 6 Months | 50
  Transplanted: BMB <50%: Survival rate at 12 Months: number analyzed (Participants) | 7
  Transplanted: BMB <50%: Survival rate at 12 Months | 42.86
  Transplanted: BMB >=50%: Survival rate at 12 Months: number analyzed (Participants) | 4
  Transplanted: BMB >=50%: Survival rate at 12 Months | 25
  Non-transplanted: BMB <50%: Survival rate at 6 Months: number analyzed (Participants) | 7
  Non-transplanted: BMB <50%: Survival rate at 6 Months | 57.14
  Non-transplanted: BMB >=50%: Survival rate at 6 Months: number analyzed (Participants) | 12
  Non-transplanted: BMB >=50%: Survival rate at 6 Months | 33.33
  Non-transplanted: BMB <50%: Survival rate at 12 Months: number analyzed (Participants) | 7
  Non-transplanted: BMB <50%: Survival rate at 12 Months | 28.57
  Non-transplanted: BMB >=50%: Survival rate at 12 Months: number analyzed (Participants) | 12
  Non-transplanted: BMB >=50%: Survival rate at 12 Months | 25

19. Secondary Outcome: Survival Rate at 6 and 12 Months in Transplanted and Non-Transplanted Elderly Participants (>65 Years)
Description: Survival rate was defined as the percentage of participants in a study or treatment group who were still alive for a certain period of time after they were diagnosed with or started treatment for a disease. In this outcome measure percentage of transplanted and non-transplanted participants greater than 65 years of age, who survived at the end of 6 months and 12 months post initiation of InO treatment are reported.
Time Frame: as for outcome 16
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 2
Percentage of participants
  Transplanted: >65 years: Survival rate at 6 Months: number analyzed (Participants) | 0
  Transplanted: >65 years: Survival rate at 12 Months: number analyzed (Participants) | 0
  Non-transplanted: >65 years: Survival rate at 6 Months | 50.0
  Non-transplanted: >65 years: Survival rate at 12 Months | 50.0

20. Secondary Outcome: Number of Participants Categorized According to Cause of Death
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 17
Participants
  Progression of disease | 4
  Relapse | 6
  Septic Shock | 2
  Veno-occlusive disease (VOD)-related multiorgan failure | 1
  VOD pneumonia | 1
  Central nervous system (CNS) relapse | 1
  Not mentioned | 2

21. Secondary Outcome: Relapse Free Survival (RFS) in All Participants and Participants With or Without Follow-up HSCT
Description: RFS was defined as time from index date to the earliest date of the following events: death, progressive disease (including objective progression, relapse from CR/CRi, treatment discontinuation due to global deterioration of health status), or the start of new induction therapy or posttherapy HSCT without achieving CR/CRi. Index date was defined as the date of initiation of the first cycle of InO. CR was defined as 5% bone marrow blasts, no evidence of disease in the bone marrow, and recovery of peripheral blood count (platelet count of >100*10^9/L and absolute neutrophil count of >1*10^9/L). CRi was defined as 5% bone marrow blasts and no evidence of disease in the bone marrow, but with incomplete recovery of peripheral blood count. Median duration of relapse free survival in all participants included those participants who had achieved CR/CRi is reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 17
Months
  All Participants | 7 [5.0 to 18.2]
  With Follow-up HSCT: number analyzed (Participants) | 9
  With Follow-up HSCT | 6 [4.8 to 10.6]
  Without Follow-up HSCT: number analyzed (Participants) | 8
  Without Follow-up HSCT | 9.5 [2.5 to 29.5]

22. Secondary Outcome: Percentage of HSCT Transplanted Participants With VOD and Percentage of HSCT Non-transplanted Participants With VOD
Description: VOD occurs when the small blood vessels in the liver are blocked.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 31
Percentage of participants
  Transplanted Participants: number analyzed (Participants) | 11
  Transplanted Participants | 45.45
  Non-transplanted Participants: number analyzed (Participants) | 20
  Non-transplanted Participants | 10

23. Secondary Outcome: Percentage of Participants With VOD in Participants Classified Per Number of Lines of Salvage Therapies
Description: VOD occurs when the small blood vessels in the liver are blocked. Salvage therapy is use of drugs after standard conventional chemotherapeutic regimens have failed to achieve remission.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. All participants reported under "Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Number; unit: Percentage of participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Percentage of participants
  First Salvage Therapy: number analyzed (Participants) | 10
  First Salvage Therapy | 20
  Second Salvage Therapy: number analyzed (Participants) | 18
  Second Salvage Therapy | 17
  Third Salvage Therapy: number analyzed (Participants) | 4
  Third Salvage Therapy | 50

24. Secondary Outcome: Percentage of Participants With VOD Classified Per High Burden and Low Burden Disease
Description: VOD occurs when the small blood vessels in the liver are blocked. Disease burden was defined using percentage of BMB. In this outcome measure low disease burden indicated BMB <50% and high disease burden indicated BMB >=50%.
Time Frame: as for outcome 1
Population: as for outcome 23
Measure: Number; unit: Percentage of participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Percentage of participants
  BMB <50%: number analyzed (Participants) | 16
  BMB <50% | 18.75
  BMB >=50%: number analyzed (Participants) | 16
  BMB >=50% | 25.00

25. Secondary Outcome: Percentage of Participants With VOD in Elderly Participants (>65 Years)
Description: VOD occurs when the small blood vessels in the liver are blocked.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 2
Percentage of participants | 50.00

26. Secondary Outcome: Number of Participants With Grade 3/4 Treatment Related Liver Toxicity (Hepatobiliary Disorder) Adverse Events (TEAEs) Following InO Initiation
Description: Treatment-related AE was any untoward medical occurrence in a participant who has received the study drug. Liver toxicity parameters included: Aspartate aminotransferase (level) >=2.5*upper limit of normal (ULN); alanine transaminase (level) >=2.5*ULN and total serum bilirubin >=1.5*ULN. Here, Grade 3 indicates severe events and Grade 4 indicates Life-threatening events where urgent intervention was required.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Participants | 12

27. Secondary Outcome: Number of Participants With Hematological Toxicities Following InO Initiation
Description: Hematological toxicities included: Febrile neutropenia= absolute neutrophil count (ANC) < 1.0*10^9 cells/L, fever >=38.5 degree C); Neutropenia= absolute granulocyte count < 1.0*10^9 cells/L; Thrombocytopenia= platelet count < 150,000 platelets per microliter.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 32
Participants | 28

28. Secondary Outcome: Number of Participants With Extramedullary Disease (EMD) or Lymphoblastic Lymphoma (LBL) Who Achieved CR or CRi
Description: Extramedullary disease was the presence of leukemic cell aggregates in the form of solid tumor outside that of bone marrow. Lymphoblastic lymphoma, was a clonal hematopoietic stem cell disorder of B or T cell origin. CR was defined as 5% bone marrow blasts, no evidence of disease in the bone marrow, and recovery of peripheral blood count (platelet count of >100*10^9/L and absolute neutrophil count of >1*10^9/L). CRi was defined as 5% bone marrow blasts and no evidence of disease in the bone marrow, but with incomplete recovery of peripheral blood count.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 2
Participants | 1

ADVERSE EVENTS:
Time Frame: From InO treatment initiation (Apr 2018) till end of follow-up (Apr 2023) [Maximum up to 61 Months]; data retrospectively collected from 08-Mar-2023 to 10-Jul-2023 (approximately 4 months of this study)
Description: AEs were reported as per participants' medical records. There was no specific medical dictionary.
Arm/Group | Inotuzumab Ozogamicin (InO)
All-Cause Mortality (participants affected / at risk) | 17/32
Serious Adverse Events (participants affected / at risk) | 19/32
Other Adverse Events (participants affected / at risk) | 28/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin (InO) (N=32)
Death (General disorders) | 17
Veno Occlusive Disease (VOD) (General disorders) | 7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin (InO) (N=32)
Aspartate aminotransferase high (Hepatobiliary disorders) | 9
Alanine aminotransferase high (Hepatobiliary disorders) | 6
Bilirubin high (Hepatobiliary disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 20
Febrile Neutropenia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT05597085/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT05597085/SAP_001.pdf